CLINICAL TRIAL: NCT03270046
Title: The Effects of An Addition of Water Enema to PEG for Colon Preparation: A Randomized Controlled Trial
Brief Title: The Effects of An Addition of Water Enema to PEG for Colon Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Somchai Leelakusolvong, Associate professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Si307/2014
Record Dates: First submitted 2017-05-03; First posted 2017-09-01 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Adenoma, Bile Duct
Keywords: Bowel preparation; CRC screening
MeSH Terms: conditions — Adenoma, Bile Duct

STUDY DESIGN:
Intervention Model Description: In this study, participants will be randomised 1:1 to water enema group or no water enema group using blocked randomization with random block sizes.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No enema group (Placebo Comparator): Consecutive participants will be randomly assigned to take a preparation regimen of 3 liter of PEG 8-16 hr. before colonoscopy without water enema.
  Before the procedure, investigators record baseline parameters. Colonoscopies underwent by experienced endoscopists and by GI fellows. During the colonoscopy, the investigators recorded video, cecal intubation and withdraw time, amount and position of polyps, rate of complete examination and complication. The video was sent to other 2 endoscopists who did not known which participant was enema to evaluate the quality of bowel cleansing by using Ottawa bowel preparation scale and Likert scale for evaluation of side effect, complication during PEG ingestion, enema and colonoscopy, and participant satisfactory.
  Interventions: Procedure: Water enema
- Water enema group (Active Comparator): Consecutive participants will be randomly assigned to take a preparation regimen of 3 liter of PEG 8-16 hr. before colonoscopy and enema with sterile water until stool was clear or patient felt discomfort but not exceed 3 liter, before colonoscopy.
  Before the procedure, investigators record baseline parameters. Colonoscopies underwent by experienced endoscopists and by GI fellows. During the colonoscopy, the investigators recorded video, cecal intubation and withdraw time, amount and position of polyps, rate of complete examination and complication.The video was sent to other 2 endoscopists who did not known which participant was enema to evaluate the quality of bowel cleansing by using Ottawa bowel preparation scale and Likert scale.
  Interventions: Procedure: Water enema

INTERVENTIONS:
Procedure: Water enema — Addition of water enema in standard PEG preparation in participants scheduled for CRC screening.

SUMMARY:
The purpose of this study is to compare the preparation quality by using Ottawa Bowel Preparation Scale between the standard PEG preparation and the addition of water enema in participants scheduled for CRC screening

DETAILED DESCRIPTION:
Background : Good bowel preparation improves the rate of polyp detection and the time of caecal intubation during colorectal cancer (CRC) screening.

Suboptimal bowel preparation can results in adenoma miss rate up to 42% (95% CI, 35-49) and advanced adenoma miss rate up to 27% (95% CI, 17-41) The European Society of Gastrointestinal Endoscopy (ESGE) Guideline recommends a split regimen of 4L of polyethylene glycol (PEG) solution (or a same-day regimen in the case of afternoon colonoscopy) for a routine bowel preparation and the delay between the last dose of bowel preparation and colonoscopy should be minimized and no longer than 4 hours.

The investigators hypothesize that the addition of water enema to the standard PEG bowel preparation could provide the better quality of bowel preparation and then result in improvement in the rate of adenoma detection among participants scheduled for CRC screening with preparation to procedure interval > 8 hr.

The purpose of this study is to compare the preparation quality using Ottawa Bowel Preparation Scale between the standard PEG preparation and the addition of water enema in participants scheduled for CRC screening. The secondary aim is to compare the effect of the standard PEG bowel preparation and the addition of water enema in terms of adenoma detection rate, the completeness of the examination, total and withdrawal time, safety and adverse events among those scheduled for CRC screening.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for CRC screening
* Bowel preparation using 3 liters of PEG solution
* Colonoscopy performed at 8-16 hours after bowel preparation

Exclusion Criteria:

* History of a failed bowel preparation
* Previous colonic surgery
* Uncontrolled underlying disease
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Bowel preparation quality using Ottawa Bowel Preparation Scale | 1 days
  Evaluate Ottawa Bowel Preparation Scale by 2 endoscopists using video record

SECONDARY OUTCOMES:
The effect of addition of water enema in standard PEG bowel preparation in terms of adenoma detection rate | 1 days
  Evaluate the adenoma detection rate compare between two groups
The effect of addition of water enema in the standard PEG bowel preparation in terms of the completeness of the examination | 1 day
  Evaluate the completeness of examination compare between two groups
The effect of addition of water enema in the standard PEG bowel preparation in terms of total and withdrawal times | 1 day
  Evaluate total and withdrawal times of colonoscopy procedures compare between two groups
The effect of addition of water enema in the standard PEG bowel preparation in terms of safety and adverse events | 3 days
  Evaluate the safety and efficacy of procedures compare between two groups

CONTACTS AND LOCATIONS:
Overall Officials: Somchai Leelakusolvong, M.D., Principal Investigator — Mahidol University

IPD SHARING:
Plan to Share IPD: No